CLINICAL TRIAL: NCT06987461
Title: Study of the Use of Non-invasive Ventilation in Bronchial Dilatation Disease (BRONCHINIV)
Brief Title: Study of the Use of Non-invasive Ventilation in Bronchial Dilatation Disease
Acronym: BRONCHINIV
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: BRONCHINIV
Record Dates: First submitted 2025-01-17; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Bronchial Dilatation Disease; Bronchectasie
Keywords: bronchial dilatation disease; Non-invasive ventilation; efficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with bronchial dilatation treated with non-invasive ventilation: Adult patients with predominantly cystic fibrosis bronchiectatic disease confirmed by tododensitometry, treated with NIV

SUMMARY:
This is a medical record data collection study. The goal of this non-interventional and retrospective study is to describe the characteristics of the population currently being monitored for bronchial dilatation who have been treated with long-term NIV. This is a study based on data from medical records.

The assessment criteria will be :

* Epidemiological characteristics of the population with bronchial dilatation on long-term NIV
* Reasons for initiation of NIV
* NIV adjustment methods

DETAILED DESCRIPTION:
Non-invasive ventilation is a treatment sometimes used for severe severe bronchial dilatation, but to date there are no studies its efficacy.

The expected results in this context are :

* a description of the characteristics of patients with severe bronchial on non-invasive ventilation (NIV)
* a better understanding, during NIV management, of the settings used, the tolerance and effectiveness of NIV in reducing exacerbations, hospital admissions and patient mortality.
* move towards better patient management

Data will be extracted from patient medical records and the PMSI.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Predominant diagnosis of bronchiectatic disease, excluding cystic fibrosis, confirmed by computed tomography
* Introduction of long-term NIV at a given point in the patient's care

Exclusion Criteria:

* Patient's opposition to participating in this study
* Cystic fibrosis
* Predominant diagnosis of COPD or asthma, traction bronchiectasis, bronchiectasis resulting from focal endobronchial lesion, sarcoidosis or active allergic bronchopulmonary aspergillosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population currently being treated for bronchial dilatation treated with long-term NIV
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
epidemiological characteristics of the population with bronchial dilation under long-term NIV | Through study completion, an average of 1 year
Reasons for placing under NIV | Through study completion, an average of 1 year
Non-invasive ventilation adjustment modalities | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
Number of acute exacerbations (according to international recommendations) after initiation of NIV | Through study completion, an average of 1 year
Stabilization of respiratory functional tests evolution of FEV1 (%, slope) of PaCO2 | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Centre Hospitalier Universitaire de Dijon, Dijon
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - Centre Hospitalier Universitaire Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No